CLINICAL TRIAL: NCT04107519
Title: Goal-Directed Resilience Training to Mitigate Chronic Pain in Former Football Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Herman A. Taylor, MD, MPH, FACC, FAHA, Director, Cardiovascular Research Institute, Morehouse School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1341910
Record Dates: First submitted 2019-06-27; First posted 2019-09-27 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Resilience; Football Players
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate GRIT (ImT) training intervention (Experimental)
  Interventions: Behavioral: Goal-Directed Resilience Training
- Delayed Training (DeT) control (No Intervention)

INTERVENTIONS:
Behavioral: Goal-Directed Resilience Training — This pilot study seeks to test the efficacy of a resilience skills training intervention for former football players who experience chronic pain. Between 20 to 48 eligible and consented participants from the Atlanta area will be identified (with a goal of 40 completing the study). They will undergo a pre-training test session and will then be randomized to either the Immediate GRIT (ImT) training intervention or the Delayed Training (DeT) control. The immediate (ImT) group will be trained for 4 weeks with 2 biweekly sessions. At the end of GRIT training they will be post-tested. The delayed (DeT) group wait during these 4 weeks and do not receive training. At the end of the 4-week waiting period, they will also be post-tested. At this point, they will be offered GRIT training for 4 weeks with 2 biweekly sessions. At the end of their training, they will be given a second post-testing. This process will then be repeated for two additional groups of 5-12 lmT and 5-12 DeT participants.
  Arms: Immediate GRIT (ImT) training intervention

SUMMARY:
The investigators propose to test a pilot study that teaches resilience skills to former football players who experience chronic pain. The purpose of this study is to see if learning resilience skills makes a difference in how former players manage chronic pain. This pilot study may advance methods to improve the well-being and quality of life of former players affected by pain.

DETAILED DESCRIPTION:
This pilot study seeks to test the efficacy of a resilience skills training intervention for former football players who experience chronic pain. Chronic pain threatens quality of life, and the culture of elite athletes is poorly adapted to the chronic condition of pain. Innovative strategies that are both culturally acceptable and effective are needed to address the needs of players who may have a reluctance to engage traditional treatment approaches.

The overarching goal is to strengthen the capacity for former football players to maintain adaptive engagement in valued activities despite chronic pain. Responding to recent findings from the Harvard Football Player Health Study (HFPHS) that identified pain as a significant challenge, we propose a pilot study that tests a resilience skills training intervention with former football players who currently experience chronic pain.

This proposed study builds on previous work conducted at Morehouse School of Medicine engaging retired professional football players and ongoing resilience intervention research involving veteran and community-based populations. The specific aim of this study is to test an intervention to decrease chronic pain and co-morbid symptoms and improve a broader adaptive level of functioning through Goal-Directed Resilience Training (GRIT) for chronic pain in a sub-sample of Atlanta-based former players.

The investigators hypothesize the following:

1. GRIT training intervention versus control training will be associated with reduced chronic pain and related symptoms of insomnia, anxiety, depression, improved emotional functions, and improved neurocognitive functions.
2. Improved self-reported physical health, quality of life, personal relationships, and personal growth will be evident for intervention versus control participants.

This pilot study has the potential to advance strategies to improve the well-being and functional status of former players impacted by pain.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Former football player between 18 - 65 of age
* Player has passed pre-selection and are referred by Harvard Football Players health study
* Potentially diverse racial & ethnic identities.

Exclusion Criteria:

* Active suicidality or suicidal intent requiring greater than outpatient level of care (Columbia Suicide Severity Rating Scale - CSSRS)
* High risk drinking of alcohol (based on scoring guidelines of AUDIT-C)
* Active psychosis (Psychosis Screener)
* Inability to participate in a small group setting (self-reported inability to regulate constructive social interaction in small group setting
* Inability to meet projected attendance requirements.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants are former professional football players; eligibility is based on self-reporting of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Focused Pain-Relevant Measures as measured by Pain Outcome Questionnaire - Short Form | Through study completion, an average of 1 year.
  Changes in pre-to-post scores for severity of pain among intervention versus control group as measured by the Pain Outcome Questionnaire. It measures severity of pain with 20 items and 6 subscales. Total range: 0-150 [20 Likert items; item range: 0-10]
  Subscales:
  Pain Intensity: 0-10 (1 item) Mobility: 0-40 (sum of 4 items) Activities of Daily Living: 0-40 (sum of 4 items) Vitality: 0 (30 minus sum of 3 items with maximum score of 10 points per item, thus 30-30=0) Negative Affect: 0-50 (sum of 5 items) Fear : 0-10 (10 minus item #18 = 0) with maximum score of 10 point for #19 Highest values = worst intensity, worst mobility, worst Activities of Daily Living, highest impaired vitality, highest negative affect, highest pain-related fear Total score: the above subscale scores are summed
Focused Pain-Relevant Measures as measured by Patient-Reported Outcomes Measurement Information System Pain Interference Short Form. | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by the Patient-Reported Outcomes Measurement Information System Pain Interference Short Form. Scale measures the extent to which pain interferes in various activities.
  Total range: 8-40 (raw score) 8 Likert items, item range = 1-5 No subscales Higher value is worse pain interference No subscales. Total raw scores is converted to t-scores.
Focused Pain-Relevant Measures as measured by Patient-Reported Outcomes Measurement Information System Sleep-Related Impairment Short Form | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Patient-Reported Outcomes Measurement Information System Sleep-Related Impairment Short Form. Measures perception of alertness, sleepiness, tiredness during waking hours.
  Total range: 8-40 raw score 8 Likert items; item range = 1-5 No subscales Higher value is worse sleep-related impairment No subscales. Total raw scores is converted to t-scores that are listed in a table in the manual.
Focused Pain-Relevant Measures as measured by Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form. Total range: 8-40 8 Likert items, item range = 1-5 No subscales Higher value is worse sleep disturbance No subscales. Total raw scores is converted to t-scores that is listed in a table in the manual
Focused Pain-Relevant Measures as measured by Pain Catastrophizing Scale (PCS) | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Pain Catastrophizing Scale (PCS). It measures fear and anxiety of pain, with 13 items Total range: 0-52 13 Likert items, item range = 0-4 No subscales Highest value = worst fear & anxiety No subscales
Focused Pain-Relevant Measures as measured by Chronic Pain Acceptance Questionnaire | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Chronic Pain Acceptance Questionnaire. It measures the acceptance of having chronic pain.
  Total range: 0-48 [8 Likert items, item range = 0-6] Subscale: Pain Willingness: 0-24 (4 items, sum of reverse scored items are: 2, 4, 7, 8) Subscale: Activity Engagement: 0-24 (4 items, sum of items 1, 3, 5, 6) Highest value=most acceptance of having chronic pain The two subscales are summed for a total score
Adaptive Functions Measures as measured by Short Form Health Survey | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Short Form Health Survey. Total range: There is no total range. All item scores of the 8 subscales are converted to scores of 0-100 according to instructions. For each subscale these are averaged, resulting in a percentage score. Highest values are the best level of functioning for subscales: physical functioning, emotional well-being, social functioning, and general health. Highest Values are also the best level of functioning for: role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, and pain.
Adaptive Functions Measures as measured by Psychological Well-being Scale | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Psychological Well-being Scale. Used 2 subscales listed below Subscale: Positive Relations with others It evaluates the extend of positive relations someone has with others. Subscale: Personal Growth It evaluates the extent to which someone values personal growth and development Total range: - the total test is not used
  Subscale range for each subscale is: 7-42 [7 Likert items; item range 1-6 for each subscale] Higher value is having or valuing highly positive relations with others, and valuing highly and seeking personal growth Positive Relations with Others: reverse scored items are 2, 3, 6. After scores are reversed, the scores for the seven items are summed.
  Personal Growth: reverse scored items are 1, 3, 5. After scores are reversed, the scores for the seven items are summed.
Adaptive Functions Measures as measured by Hedonic and Eudaimonic Motives for Activities | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Hedonic and Eudaimonic Motives for Activities. This scale assesses the extent to which someone values happiness and pleasure versus seeking self-growth.
  Total range: 9-63 [9 Likert items, item range 1-7] Hedonia subscale: 5-35 Eudaimonia subscale: 4-28 Hedonia subscale: higher value means valuing and seeking happiness and pleasure Eudaimonia subscale: higher value means seeking self-development and being the best a person can be Subscales are not combined but sand alone. Hedonia subscale: consists of 5 items: 1, 4, 6, 7, 9. To obtain a score, item scores are summed Eudaimonia subscale: consists of 4 items: 2, 3, 5, 8. To obtain a score, item scores are summed.
Adaptive Functions Measures as measured by Patient Health Questionnaire | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Patient Health Questionnaire. This scale measures the extent to which someone feels depressed Total range: 0-27 [9 Likert items, item range 0-3] No subscale High value is worse depression No subscales To obtain a total score, the 9 item scores are summed
Adaptive Functions Measures as measured by Generalized Anxiety Disorder Scale | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Generalized Anxiety Disorder Scale This scale measures the extent to which someone feels anxious or fearful Total range: 0-21 [7 Likert items, item range 0-3] No subscale Higher value is worse or high level of anxiety No subscales To obtain a total score, the 7 item scores are summed
Adaptive Functions Measures as measured by Adverse Childhood Experience Questionnaire | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Adverse Childhood Experience Questionnaire This measures the extent to which someone has experienced adversities in poor treatment, family disruption, abuse, etc. during childhood Total range: 0-10 [10 Yes No questions, Yes=1, No=0] No subscales Higher value is higher and more experience of childhood adversity and abuse No subscales To obtain a total score, the 10 items are summed
Neurocognitive Measures as measured by Delis-Kaplan Executive Function System | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Delis-Kaplan Executive Function System. This battery measures neuropsychological executive functions or complex aspects of reasoning. Individual test scores are frequency counts of correct responses or length of time on the items of subscale, and frequency of errors. Verbal Fluency Test = higher value is better verbal fluency Color-Word Interference Test = higher score on time taken to complete is worse performance. Verbal Fluency Test consists of 4 sub-tests that stand alone: Letter Fluency, Category Fluency, Category Switching Total Correct, Category Switching Accuracy.
Neurocognitive Measures as measured by Repeatable Battery for the Assessment of Neuropsychological Status | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Repeatable Battery for the Assessment of Neuropsychological Status Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) This battery assesses a range of neurocognitive functions, including learning, episodic memory, working memory, complex attention.
  Total range: There is no total range, just individual test ranges. Individual test range: individual test scores are frequency counts of correct responses or length of time taken for one subtest. There is no range.
  Higher correct performance scores are better. Higher scores for taking more time are worse.
  Several tests from this battery are used. These stand alone:
  List Learning, Story Memory, Digit Span, Coding, List Recall, List Recognition, Story Recall. For each test the raw performance is summed and recorded and a scaled score that is found in the manual is also recorded.
Neurocognitive Measures as measured by Neuropsychological Assessment Battery | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group as measured by Neuropsychological Assessment Battery This is a comprehensive battery that assesses a wide range of neurocognitive functions.
  Total range: There is no total range, just individual test range. Individual test range: individual test range is the frequency counts of correct responses. Also counted are perseverative errors. There is no range.
  Higher value of summed correct responses is better. Higher value of perseverative errors is worse. One sub-test is used from this battery: Word Generation. It stands alone. Total sub-test score is the number of correct words generated. Perseverative errors are total number of errors committed.
Resilience Resources for the Unpredictability of Chronic Pain | Through study completion, an average of 1 year.
  Changes in pre-to-post scores among intervention versus control group. This scale consists of two subscales that measure the unpredictability of pain and resilient responses to pain comprised of engagement in activities, cultivating social relations, and pursuing self-growth.
  Unpredictability of Chronic Pain covers inability to predict when the person will be in pain, how long it will last, how much person could not plan his activities, how much it interfered in relationships. The size of the score on this subscale will indicate the size of unpredictability of pain Resilience Resources cover three domains: (1) engagement with interest, curiosity, appreciation, noticing beauty in activities despite pain (2) pursuing relationships in showing empathy, helping, friendship, compassion (3) self-growth to pursue excellence, to grow as a person, to learn new skills to improve oneself.
Physical Functions Measure | Through study completion, an average of 1 year.
  Time Measure of Walking. The Six minute walk test is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism.

SECONDARY OUTCOMES:
Physiologic measurement of Blood Pressure (BP) | Through study completion, an average of 1 year.
  Changes in pre-to-post scores for blood pressure among intervention versus control group. The auscultatory method of BP measurement with a properly calibrated and validated instrument will be used. Patients will be seated quietly for at least 5 minutes in a chair rather than on an examination table, with feet on the floor and arm supported at heart level. An appropriate-sized cuff (cuff bladder encircling at least 80% of the arm) will be used to ensure accuracy. At least 2 measurements will be made. Systolic BP is the point at which the first of 2 or more sounds is heard (phase 1) and diastolic BP is the point before the disappearance of sounds (phase 5).

CONTACTS AND LOCATIONS:
Overall Officials: Herman Taylor, MD, MPH, Principal Investigator — Cardiovascular Research Institute
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04107519/Prot_SAP_000.pdf